CLINICAL TRIAL: NCT06735352
Title: Effect of Vırtual Realıty Glasses on Mıld Cognıtıve Impaırment in Elderly: A Randomızed Controlled Study
Brief Title: Effect of Vırtual Realıty Glasses on Mıld Cognıtıve Impaırment in Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Buket DAŞTAN, Assist. Prof. Dr., Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: RCS15102024
Record Dates: First submitted 2024-12-05; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Mild Cognitive Impairment (MCI)
Keywords: elderly; virtual reality; mild cognitive impairment; nursing
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): No intervention was made to the elderly in this group.
- virtual reality group (Experimental): Evaluated the effect of using virtual reality in elderly people with mild cognitive impairment.
  Interventions: Other: virtual reality intervention

INTERVENTIONS:
Other: virtual reality intervention — Evaluated the effect of virtual reality use in elderly people with mild cognitive impairment compared to a control group.
  Arms: virtual reality group

SUMMARY:
This study was conducted in a randomized controlled manner to investigate the effect of VR glasses on mild cognitive impairment in the elderly. The main questions the study aimed to answer are:

• Will VR improve mild cognitive impairment in the elderly? The researchers used a control group to compare the effect of VR on mild cognitive impairment.

Participants:

* Before starting the study, the elderly were given the necessary forms and information.
* The elderly were shown virtual reality videos with VR glasses 3 days a week for 4 weeks.
* The control group did not watch any videos, and the post-test forms were filled out again for both groups at the end of 4 weeks.

DETAILED DESCRIPTION:
The elderly population rate is rapidly increasing in the world and in our country. According to the World Health Organization (WHO) data, the elderly population aged 60 and over, which was 1 billion in 2019, is expected to increase to 1.4 billion in 2030 and 2.1 billion in 2050. In our country, the elderly population, which was 6 million in 2016, reached more than 8 million in 2023. (WHO 2021, TÜİK 2024). As life expectancy continues to increase, the number of elderly people who cannot live independently and need assistance due to cognitive decline is rapidly increasing worldwide (Díaz-Pérez &, Flórez-Lozano, 2018; Huang & Yang, 2022). Dementia is a collective name for a heterogeneous group of chronic neurodegenerative diseases characterized by progressive impairment of behavior and cognitive function (Aruanno & Garzotto, 2019; D'Cunha et al., 2019). Mild Cognitive Impairment (MCI) is an intermediate stage of cognitive change between normal aging and dementia; the distinction between MCI and dementia is determined by the severity of cognitive decline leading to functional impairment. MCI, also known as the "symptomatic predementia stage," causes mild deterioration in cognitive function without significant loss of independent functional abilities, social and occupational functioning in individuals (Kim et al., 2019). MCI is defined as a condition in which individuals experience memory loss greater than expected for their age but do not meet the criteria for dementia. This is a less severe degree of cognitive impairment compared to dementia and is classified as Mild Cognitive Impairment in the DSM-5. However, the capacity for independence in activities of daily living and instrumental activities of daily living is preserved, unlike diseases such as dementia (Oliveira et al., 2021). According to WHO, there are approximately 55 million people with dementia worldwide; this number is expected to increase to 75 million by 2030 and approximately 135 million by 2050 (WHO, 2023). However, individuals with MCI typically have a higher risk of dementia than individuals of the same age without MCI (Petersen et al., 2018; Aruanno & Garzotto, 2019; Kim et al., 2019). Although pharmacological interventions are recommended for the treatment of dementia types and MCI, polypharmacy in the elderly population can cause side effects. Therefore, new and effective non-pharmacological treatments are needed (Huang & Yang 2022). Updated practice guidelines have indicated that exercise and cognitive interventions may be beneficial for improving cognitive functions in patients with MCI (Kim et al., 2019). Participation in stimulation of mental activities in older ages may be a protective factor against cognitive decline and possibly reduce the risk of developing dementia (Manera et al., 2016). Virtual reality (VR) is a new technology used for the rehabilitation of cognitive and motor functions (Tieri et al., 2018). VR is defined as a real or imaginary three-dimensional environment of computer simulation that allows its users to experience the feeling of being in a different physical place (D'Cunha et al., 2019). VR is a new branch of computer technologies that has recently been proposed for use in the field of neuropsychology. VR is a high-level computer interface that includes real-time simulation and interactions through multiple sensory channels, based on various perception components of psychophysics, primarily visual, tactile and kinesthetic perceptual sensations. The use of VR systems offers the opportunity to simulate immersive and interactive real-life scenarios to create a sense of "being there" (Zhu et al., 2021). The use of VR systems for disease treatment has already been investigated in various fields such as brain injury, post-stroke intervention, and musculoskeletal recovery. VR environments have also been used for neuropsychological assessment and problems such as phobias, stress, anxiety, exercise, and memory problems (Luque-Moreno et al., 2021; Manera et al., 2016). It has been reported that the use of VR for both stimulation and relaxation in people with cognitive decline reduces stress. These studies suggest that virtual reality can be used as a promising tool in many therapeutic and rehabilitation areas in MCI and dementia and have attracted the attention of researchers (Manera et al., 2016). Therefore, this study aimed to determine the effect of VR intervention on MCI in elderly individuals.

ELIGIBILITY:
Inclusion Criteria:

* The study included elderly individuals who were over the age of 65,
* Diagnosed with MCI by a neurologist,
* Having a Standard Mini-Mental Statement (MMSE) score between 18 and 23,
* Having a Montreal Cognitive Assessment Scale (MOCA) score below 21,
* Able to communicate verbally,
* Agreeing to participate in the study.

Exclusion Criteria:

* The study excluded those with a history of stroke or epilepsy,
* Those with other suspected degenerative diseases or diagnosed severe psychiatric illnesses,
* Those with head trauma, thyroid disorders or other medical abnormalities that could impair cognitive function.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Elderly Information Form | 4 week
  The study includes questions to determine the age, gender, marital status, education level and chronic disease status of elderly individuals.
Mini-Mental State Examination | 4 week
  The MMSE, which provides assessment of cognitive status, was developed by Folstein and colleagues in 1975 and is the most commonly used and easily administered test in dementia screening (Folstein, 1975). Its validity and reliability in the diagnosis of mild dementia for the Turkish population was performed by Güngen and colleagues (Güngen 2002). The mini mental test is grouped under five main headings: orientation (10 points), recording memory (3 points), attention and calculation (5 points), recall (3 points) and language (9 points). The scale is evaluated out of a total of 30 points and has two different types for the educated and the uneducated. Traditionally, scores between 24 and 30 are considered normal. A score below 24 indicates cognitive impairment. A score between 18-23 points is considered mild dementia, 12-17 points is considered moderate dementia and 12 points below is considered severe dementia.
Montreal Cognitive Assessment Scale | 4 week
  It is a screening scale developed specifically to evaluate the early stages of cognitive impairment. The scale evaluates attention and concentration, executive functions, memory, language, visual and spatial skills, abstract thinking, calculation and orientation functions. The test takes approximately 10 minutes. The visual structuring skills test is worth 5 points, the attention test is worth 6 points, the language (naming) test is worth 6 points, the abstract thinking test is worth 2 points, the delayed recall is worth 5 points and the orientation test is worth 6 points. Patients with 21 points and above out of 30 points are considered cognitively normal.

CONTACTS AND LOCATIONS:
Overall Officials: Buket DAŞTAN, Ph.D, Principal Investigator — Karadeniz Tecnic University
Locations (1):
- Bayburt State Hospital, Bayburt, Centre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
I'll decide later